CLINICAL TRIAL: NCT03895957
Title: VR Mind™ and VR Mind +™ Intervention - Randomized, Open Label, Single Masking, Parallel Group Clinical Trial
Brief Title: VR Mind and VR Mind+ Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomorrow Sp. z o.o. (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRR/POIR.01.01.01-00-0636
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2019-03

CONDITIONS: Social Phobia
Keywords: virtual reality; social phobia; vret; virtual reality exposure therapy
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: VR Mind+ (Experimental): Virtual Reality Exposure Therapy VR Mind+
  Interventions: Behavioral: Virtual Reality Exposure Therapy VR Mind+
- Group 2: VR Mind (Experimental): Virtual Reality Exposure Therapy VR Mind
  Interventions: Behavioral: Virtual Reality Exposure Therapy VR Mind
- Control group: CBT (Active Comparator): Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy VR Mind+ — Virtual Reality Exposure Self-Therapy led by a participant
  Arms: Group 1: VR Mind+
Behavioral: Virtual Reality Exposure Therapy VR Mind — Treatment with Virtual Reality Exposure Therapy led by a therapist
  Arms: Group 2: VR Mind
Behavioral: Cognitive Behavioral Therapy — Standard treatment for social phobia led by a therapist
  Arms: Control group: CBT

SUMMARY:
The aim of the study is to assess the safety and efficacy of VR Mind and VR Mind + interventions.

DETAILED DESCRIPTION:
In this study, investigators will test the software developed by Tomorrow Sp. z o. o., named VR Mind and VR Mind+. The software utilizes the concept of virtual reality exposure therapy to treat social anxiety disorder. The aim of the study is to assess the safety and efficacy of VR Mind and VR Mind + interventions.

The research consists of fourteen sessions. The first and the last session will be dedicated to participant assessment. Subsequent sessions 2-13 will be performed according to the therapy protocol for each arm. Control group of participants (active comparative arm) will receive standard treatment for social anxiety disorder - cognitive behavioral therapy based on the protocol developed by the Principal Investigator [protocol adapted from the approach of Clark and Wells (Mayo-Wilson, Dias, Mavranezouli, 2014)]. Experimental group 1 will receive cognitive behavioral therapy with exposure in virtual environment. Experimental group 1 and control group were designed to be as similar as possible, with the exception of the modality for the delivery of exposure. All treatment session will be led by licensed therapist.

Participants of the experimental group 2 will independently conducts the self-therapy process. The intervention will consist of 12 therapeutic sessions. At each of the 12 sessions, the participant will selects a specific scenario of social situations that arouse fear (e.g. public speaking, job interview or other situations from everyday life).

Because of the risk of simulator sickness (e.g., headaches, nausea), exposure trials will last no longer than 20 minutes for each session.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed DSM-IV-TR criteria for Social Anxiety Disorder (SAD).
* Signing informed consent
* Unchanged doses of psychotropic medications within 3 months prior to baseline assessment and no change is anticipated

Exclusion Criteria:

* occurrence of SAD symptoms inconsistent with DSM-IV-TR criteria and with psychiatric interview (SCID-I; Structured Clinical Interview)
* psychosis,
* bipolar disorder,
* mental retardation
* pregnancy,
* drug addiction,
* alcohol addiction,
* psychoactive substances addiction,
* participating in the experimental session while intoxicated
* (current) neurological treatment of chronic disease of central nervous system,
* epilepsy,
* paroxysmal vertigo,
* presence of suicidal thoughts, tendencies or attempts,
* participant is taking drugs from benzodiazepine group, other sedatives, narcotic drugs
* current CBT treatment for Social Anxiety Disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy: Liebowitz Social Anxiety Scale - Liebowitz Social Anxiety Scale (LSAS; Liebowitz, 1987) | change from baseline: Pre-treatment at session 1, to session 9 (5 weeks) and to post-treatment at session 14 (7 weeks)
  The scale is composed of 24 items, depicting various social situations. For each item, participants assess their fear (from 1 - "No fear" to 4 - "Severe") and avoidance (from 1 - "Never" to 4 - "Usually"). LSAS has 3 scores, summing the results for particular items - fear (0-72), avoidance (0-72) and total score (0-144).
Safety: Occurrence and severity of Simulator Sickness - Simulator Sickness Questionnaire (SSQ; Kennedy, Lane, Berbaum, Lilienthal, 1993) | Change from session to session with virtual reality exposure: at session 1, session 7 (4 weeks), session 8 (4 weeks), session 10 (5 weeks), session 11 (6 weeks) and session 12 (6 weeks)
  Simulator sickness is expected adverse effect of the VR.Total SSQ score equal to or higher than 10 will be used as a preliminary cut-off for simulator sickness (Balk et al., 2013). Individual scores will be corrected for baseline (pre-VR) symptom severity. Only items with a pre-VR - post-VR increase will contribute to a final SSQ score. All post-intervention SSQ scores >10 will be analyzed further for its association with study drop-outs and other intervention required. The adverse effect will be classified as:
  * mild (no intervention required),
  * moderate (any intervention needed, e.g. session termination),
  * severe (hospitalization required),
  * life-threatening / death.
  Some of the symptoms of anxiety may produce similar side effects as a simulator sickness. The results obtained in this case will be false positive. Therefore assessment of side effects for each case will be verified if the increase in SSQ score was triggered by rapid relapse of phobia symptoms.

SECONDARY OUTCOMES:
Clinical Global Impression | Pre-treatment at session 1
  Clinical Global Impression (CGI; Guy, 1976) - is a single item, 7 point scale used by clinicians to assess the severity of illness, where 1 is labeled as "Normal, not at all ill" and 7 is labeled as "Among the most extremely ill patients".
Clinician Global Impressions of Improvement | Post-treatment, approximately 7 weeks after initial session
  Global measure of change in severity of symptoms, ranging from 1 labeled as " Very much improved" to 7 labeled as "Very much worse".
Patient Global Impression | Pre-treatment at session 1
  Patient Global Impression - is a single item, 4 point scale used by patients to assess their impression of severity of their illness and quality of their functioning in everyday life, where 1 is labeled as "Normal" and 4 is labeled as "Severe".
Patient Global Impressions of Improvement | Post-treatment, approximately 7 weeks after initial session
  Global measure of change in severity of symptoms, where 1 is labeled as "No change" and 7 is labeled as " Very much improved ".
Beck Depression Inventory | Pre-treatment at session 1 to post-treatment at session 14 (7 weeks)
  A 21-question multiple-choice self-report inventory for measuring the severity of depression. Each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original:
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression

OTHER OUTCOMES:
Subjective Units of Distress | Change from session to session with virtual reality exposure during the course of six weeks
  Subjective Units of Distress (SUD) SUD is a subjective measure of perceived fear in certain situation. The scale range is from 0 ("Totally relaxed) to 100 ("Highest distress/fear/anxiety/discomfort that you have ever felt").

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Mierzejewski, prof., Study Chair — Scientific Council; Przemysław Bieńkowski, prof., Study Director — Scientific Council; Tadeusz Parnowski, prof., Study Director — Scientific Council; Sławomir Murawiec, PH.D., Study Director — Scientific Council; Izabela Stefaniak, M.D., Principal Investigator — Scientific Council
Locations (2):
- Poland (2):
  - Tomorrow Sp. z o. o., Warsaw
  - Gabinet Psychoterapii, Warsaw

IPD SHARING:
Plan to Share IPD: No